CLINICAL TRIAL: NCT06273488
Title: The Role of Auricular Acupoint Diagnosis and Therapy in Enhanced Recovery After Surgery of Total Knee Arthroplasty Based on Real World Study
Brief Title: The Role of Auricular Point Diagnosis and Treatment in ERAS During TKA
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Qindong Mi, research assistant, Peking Union Medical College
Other Study IDs: EXZL20240002
Record Dates: First submitted 2024-01-31; First posted 2024-02-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Auriculotherapy; Arthroplasty, Replacement, Knee; Enhanced Recovery After Surgery
MeSH Terms: interventions — Auriculotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Auriculotherapy intervention group
  Interventions: Other: Auriculotherapy
- Control group

INTERVENTIONS:
Other: Auriculotherapy — Treatment of pain, drug addictions, or other ailments by stimulating the various points on the external ear (EAR AURICLES). It is based on the ancient Chinese practices of EAR ACUPUNCTURE, but sometimes magnets and other modes of stimulation are used.
  Groups: Auriculotherapy intervention group

SUMMARY:
To further improve the surgical outcomes of patients undergoing total knee arthroplasty (TKA). This study aims to use ear acupoint therapy to address the following clinical issues: 1 The degree of postoperative inflammation and edema in the patient; 2. Patient pain; 3. Patient functional recovery. 4. Surgical scar repair for patients; 5. Patient perioperative anxiety and postoperative satisfaction. Exploring the safety and effectiveness of ear acupoint therapy in the postoperative application of TKA, leveraging the advantages of suitable traditional Chinese medicine techniques in simplicity, convenience, effectiveness, and cost-effectiveness, and further improving the ERAS Chinese and Western medicine collaborative plan for TKA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years old, no gender limit;
2. Meet the late diagnostic criteria for knee osteoarthritis and meet the surgical indications for TKA;
3. The patient's auricles of both ears are intact
4. The subject/guardian makes it clear that the patient will choose to go to a medical consortium hospital for standardized medical treatment after surgery.

   Repeat treatment.
5. Subjects/guardians can understand the purpose of the trial and show sufficient compliance with the trial protocol,and signed the informed consent form (ICF).

Exclusion Criteria:

1. Suffering from severe arrhythmia, heart failure, chronic obstructive pulmonary disease, epilepsy, mental illness sick;
2. The patient's ears are damaged, red, swollen, bleeding, infected, etc. and have contraindications that are not suitable for auricular acupoint diagnosis and treatment.
3. Patients with knee varus >15° or valgus before surgery;
4. Other circumstances in which the researcher deems it inappropriate to participate in this clinical trial.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo TKA to treat KOA in the Department of Orthopedics of Peking Union Medical College Hospital from March to December 2024.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in Range of motion(△AROM) | The change in AROM from postoperative day 1 to day 4 (measured by trained personnel to optimize accuracy) was used as the primary outcome measure.
  Active range of motion (AROM) is defined as the degree of knee flexion achieved without assistance. It is closely related to lower limb pain, kinesiophobia and swelling, and better reflects the early functional recovery of the knee joint after surgery.

SECONDARY OUTCOMES:
Facial Visual Analog Scale (VAS-F) | preoperatively and on postoperative Days 1-4, 7 and 14 during early rehabilitation exercise
  The Face Visual Analogue Scale (VAS-F) is a tool used to assess subjective experiences such as pain, discomfort, or emotional states. It utilizes a visual scale with facial expressions ranging from "very happy" to "very sad" or "no pain" to "worst pain imaginable," allowing patients to self-report their feelings or symptoms.
  Measurement Procedure:
  Scale Presentation:The patient is presented with a horizontal line (typically 10 cm in length) accompanied by a series of facial expressions at each end.On the left end, a "very happy" or "no pain" face is displayed, representing the best possible condition (score: 0).On the right end, a "very sad" or "worst pain imaginable" face is displayed, representing the worst possible condition (score: 10).
Self-Assessment Survey for Anxiety（SAS） | Within 3 days before surgery
  The SAS score is a tool used to assess an individual's anxiety status, typically used in adults and adolescents. The cut-off value of the standard score is 50 points. A score below this indicates no anxiety problems, while a score above this may indicate varying degrees of anxiety problems.
  According to the increase in anxiety level, SAS scores can be divided into mild (50-59 points), moderate (60-69 points), and severe (over 70 points) anxiety. This study evaluated the perioperative anxiety of patients using this scale.
Acupoint electrical measurement value(AE) | Within 3 days before surgery and 1 month after surgery
  Measure the electrical measurement values of acupoints in corresponding parts of the body through a meridian analyzer.
Dosage of painkillers | Within 1 months after surgery
  Including the dosage of non steroidal anti-inflammatory drugs and the number of times the pain pump is pressed.
Hospital stay | Within 1 months after surgery
  Including wish days during acute and recovery periods
HSS knee joint scoring | postoperative Days 7 and 14
  The HSS knee joint scoring system is a scoring system proposed by the Hospital for Special Surgery in the United States in 1976 to evaluate preoperative and postoperative knee joint function. It mainly includes six aspects: pain, function, joint range of motion, muscle strength, knee flexion deformity, knee instability, etc., with a maximum score of 100 points. The clinical efficacy classification is excellent>85, good 70-84, medium 60-69, and poor<59. Use this scale to comprehensively evaluate the postoperative functional recovery of the knee joint.
Thigh circumference(knee joint circumference) | postoperative days 1-4, and 14
  The leg circumference measurement method is mainly used to evaluate the swelling of lower limbs after TKA.
Kine siphobia (TSK) score | postoperative days 1-4, 7 and 14
  Use this scale to evaluate patients' postoperative kinesiology. This scale has 17 items in total, with a total score of 17 to 68 points. A score of >37 can be diagnosed as kinesiphobia. The higher the score, the higher the degree of kinesiphobia after TKA.
C-reactive protein (CRP) | Within 3 days before surgery and 4 days after surgery
  This indicator was collected through review of medical records
Erythrocyte Sedimentation Rate(ESR) | Within 3 days before surgery and 4 days after surgery
  This indicator was collected through review of medical records.
Postoperative satisfaction | 1 month after surgery
  Investigate patients' satisfaction with auricular acupuncture diagnosis and treatment mainly through telephone follow-up.
Expenses during hospitalization | Within 3 days after the patient leaves the surgical hospital
  This indicator was collected through review of medical records
Demand rate and satisfaction rate of auricular point diagnosis and treatment | 1 month after surgery
  The demand rate calculation formula is the total number of patients who require ear acupuncture treatment/included in this study, while the satisfaction rate calculation formula is the final patient who provides ear acupuncture treatment/patient who requires ear acupuncture treatment.
Adverse events related to auricular acupuncture diagnosis and treatment | Within 1 month after surgery
  Adverse events related to auricular acupuncture diagnosis and treatment
Affected limb drainage volume | Within 4 days after surgery
  This indicator was collected through review of medical records
Preoperative Anxiety Scale (PAS-7) score | 24±2h after the start of AP or first visit, 12±2h before surgery, and 2 h before surgery.
  This scale assesses some of the patient's conditions related to surgery, and then selects the appropriate option among the 5 options based on the actual situation during the few days of hospitalization, and circles the corresponding number. The higher the score, the more severe the patient's preoperative anxiety.This scale consists of 7 questions, with a total score of 28 points. The higher the score, the more severe the patient's preoperative anxiety level is
patient-controlled analgesia (PCA) pressing times | postoperative Days 1-4
  This indicator was collected through review of medical records
Modified Pittsburgh Sleep Quality Index (M-PSQI) | 24±2h after the start of AP or first visit , 12±2h before surgery, and 72±2h post-operatively.
  To accommodate the short treatment duration and unique ward environment of hospitalized patients, this study modified the Pittsburgh Sleep Quality Index (PSQI) to develop an adapted version (M-PSQI) for short-term sleep assessment. The scale consists of 24 items (19 self-rated + 5 caregiver-rated), with scoring based on the 19 self-rated items, which assess the following dimensions:
  1. Sleep Process Metrics: Sleep latency, total sleep duration, wake time
  2. Sleep Disturbance Manifestations: Difficulty falling asleep, nocturnal awakening frequency, environmental/physiological sleep disruptions
  3. Subjective Sleep Quality: Patients' overall evaluation of sleep quality
  4. Medication Use: Frequency of sedative-hypnotic drug use
  5. Daytime Functional Impairment: Difficulty maintaining wakefulness, reduced task performance efficiency The scale adopts a 7-factor structure, with each factor scored on a 0-3 scale. The total score ranges from 0 to 21, with higher scores indicating more severe sleep
Patient Satisfaction with Pre-operative Preparation Assessed with the Visual Analogue Scale (VAS-Satisfaction) | 2 h before surgery
  The Visual Analogue Scale for Satisfaction (VAS-Satisfaction) is a simple, validated tool used to measure a patient's subjective satisfaction with their pre-operative preparation. It consists of a 100-mm horizontal line anchored by two extreme statements: Left anchor (0 mm): "Not satisfied at all"; Right anchor (100 mm): "Completely satisfied".
  The patient marks a point on the line corresponding to their level of satisfaction with the pre-operative process (This includes the information provided before surgery, the attitude of the medical staff, the arrangement of the preoperative process, and the overall experience of preoperative preparation). The score is quantified by measuring the distance (in mm) from the left anchor to the patient's mark, yielding a numerical value between 0 (lowest satisfaction) and 100 (highest satisfaction).
AROM | AROM of the knee joint was assessed by trained personnel preoperatively and on postoperative days 1-4, 7, and 14 repectively to observe the recovery trend of AROM after surgery
5-point Verbal Rating Scale (VRS-5) | postoperative day 30
  The 5-point Verbal Rating Scale (VRS-5) is a simple method for assessing pain intensity, typically involving the following steps:
  Ask the patient to describe their pain using one of the following five predefined categories:
  0: No pain - No discomfort or pain at all.
  1. Mild pain - Pain is noticeable but easily tolerated.
  2. Moderate pain - Pain is more pronounced and may interfere with daily activities.
  3. Severe pain - Pain is intense and difficult to tolerate, significantly impacting daily life.
  4. Very severe pain - Pain is excruciating and unbearable, often requiring immediate relief.
  Record the patient's response as a numerical value (0 to 4) based on their description.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No